





## **COGNITION AND FLOW STUDY PARTICIPANT CONSENT FORM (PATIENT)**

| 200 | Trust Patient Study ID Number: | Please initial |
|---|---|---|
| Date | I confirm that I have read and understand the Information Leaflet ( <i>Version 4, ed 08/01/2019</i> ) for the above study, and have had the opportunity to ask questions and e had these answered satisfactorily. | |
| | I understand that my participation is voluntary and that I am free to withdraw at any e, without giving reason, without my medical care or legal rights being affected. | |
| rese | I understand that if I decide to withdraw prior to the completion of the study, the earch team would like to keep all the health information and data that has n collected so far for the final analysis, and I am granting permission for this. | |
| cons | If I lose the ability to make decisions for myself during the study I would like to be sidered to remain in the study, if my relative, carer or friends felt it was appropriate for to do so. Please circle yes or no. | |
| Info | I understand that Lumosity© will monitor my use of the brain training program and provide rmation to the research team about frequency and duration of use. These data will be nymised and no personal information will be shared. | |
| | I understand that my GP will be informed about my participation in this study, and by ing this consent form I am granting permission for this. | |
| of p | I understand that if there are any health concerns identified as a result articipation in this study, my GP will be informed to investigate this further and by signing consent form I am granting permission for this. | |
| stuc<br>NHS | I understand that relevant sections of my medical notes and/or data collected during the dy, may be looked at by responsible individuals from the study team, the sponsor, a Trust or from regulatory authorities, where it is relevant to taking part in this research. The permission for these individuals to have access to my records. | |
| conf<br>oth | I understand that any information I provide during this study will remain fidential unless there are any serious concerns about my safety or the safety of ers. I understand that the researcher will firstly speak to me before making any losures. | |
| | OPTIONAL I agree to take part in a focus group with the other participants, or nterview. | |
| 11. | OPTIONAL I agree to the interviews / focus groups being audio-recorded. | |
| | I understand that I can withdraw my interview/focus group data from the study at any a until it is anonymously transcribed. | |

| 13. OPTIONAL I give permission for Quoted directly in published reports results will be anonymised, and all p | s. I understand that anything | which is included in the final |
|---|---|---|
| any published reports. | | |
| 14. I would like a lay summary of the results of the study sent to me by <u>post</u> or <u>email</u> (please | | |
| circle) at the end of the study . | | |
| 15. I agree to take part in the above | e study. | |
| Participant Name: | Date: | Signature: |
| Researcher: | Date: | Signature: |
| (File: 1 for participant, 1 for research | her, 1 for hospital notes) | |